CLINICAL TRIAL: NCT00071916
Title: African American Response to Therapy for Hepatitis C
Brief Title: Racial Difference in HCV/Host Interactions
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jaquelyn Fleckenstein, University of Tennessee
Other Study IDs: 00-091
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2010-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C, African Americans, ribavirin
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood. No liver biopsies will be performed specifically for inclusion into the tissue repository. Only slides or paraffin tissue blocks of previously performed liver biopsies will be included in the tissue repository.

GROUPS / COHORTS (2):
- African American: Adult African American participants with compensated chronic hepatitis C who have not been previously been treated with interferon and/or ribavirin.
- Caucasian: Caucasian participants with compensated chronic hepatitis C who have not been previously been treated with interferon and/or ribavirin.

SUMMARY:
The purpose of this study is to evaluate a group of African Americans and Caucasians with hepatitis C virus (HCV), compare their response rates to combination treatment with pegylated interferon alfa-2b and ribavirin, and identify possible causes for racial differences in response to therapy. The study will enroll a total of 260 participants, age 18 or older, over a 10 period. In the next 5 years 132 subjects will be studied locally, including 112 African Americans and 20 Caucasians. Participants will be recruited from the clinical practices of the hepatologists (liver doctors) at the University of Tennessee Health Science Center and will also be selected from referrals at local hepatology clinics and the Memphis VA Hospital. Volunteers will be treated with pegylated interferon alfa-2b injections once weekly and oral ribavirin 2 times a day for up to 72 weeks. Study procedures include multiple blood draws. Participants may be involved in study related procedures for up to 72 weeks.

DETAILED DESCRIPTION:
The University of Tennessee Health Science Center (UTHSC) Memphis Hepatitis C Cooperative Research Center was established in 2000 to support clinical and basic research in understanding the basis for chronic disease in hepatitis C (HCV) infection and response to therapy in clinically infected patients. The primary research goal is to understand why African American (AA) patients with chronic hepatitis C are more susceptible to chronic infection and why their response rate to combination therapy is only 50 percent or less of that for non AA patients. The present study will support this ongoing work by continuing to provide clinical samples from patients with chronic hepatitis C who are undergoing treatment. The specific aims for the 2005-2010 Hepatitis C Cooperative Research Center are: to determine how human leukocyte antigen (HLA) class II-dependent immune regulation and T cell specificities affect differences in immune responses to HCV and response to therapy in AA patients compared to non AA patients; to determine if there is a difference in interferon-induced signaling between patients that respond to therapy and those that do not; and to measure and compare the sustained virologic response to standard treatment for hepatitis C between AA and non AA patients. Researchers plan to continue enrollment of patients to the "African American Response to Therapy for Hepatitis C" study (112 African American patients and 20 Caucasian patients) in order to meet the current specific aims. Participants will include adult African American and Caucasian patients with compensated chronic hepatitis C who have not been previously treated with interferon and/or ribavirin. Patients meeting the entry criteria will be enrolled. The total number of patients to be enrolled is 260 over a 10-year period. In the next 5 years 132 subjects (112 African American, 20 Caucasian) will be studied locally. Patients will be recruited primarily from the clinical practices of the hepatologists at UTHSC. Patients will also be selected from referrals at local Gastroenterology Hepatology clinics and the Memphis Department of Veterans Affairs (VA) Hospital. Patients will be treated with weight based pegylated interferon alfa-2b once weekly and weight based ribavirin twice a day. Duration of treatment with both pegylated interferon alfa-2b and ribavirin will be for up to 72 weeks. Treatment will be discontinued at 24 weeks if there is persistent viremia and the patient wishes to discontinue therapy. Ribavirin will be administered orally at a dose of 13 +/- 2 mg/kg per day twice daily, with 200 mg capsules. Pegylated interferon alpha-2b will be administered by the subcutaneous route.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male or female, African-American or Caucasian, age 18 or older.
* Serum positive for hepatitis C virus by Polymerase Chain Reaction (PCR) or other assays [e.g. Deoxyribonucleic acid, (BDNA)].
* Liver biopsy prior to entry to this protocol with a pathology report confirming that the histological diagnosis is consistent with chronic hepatitis.
* Compensated liver disease with the following laboratory parameters at the Entry visit:
* Hemoglobin values of greater than or equal to 12 mg/dL
* Neutrophil count greater than or equal to 1,200/mm^3
* Platelets greater than or equal to 60,000/mm
* Albumin > 3.0 g/dL or within 20 percent of lower limit of normal (LLN)
* Serum creatinine less than or equal to 1.5 mg/dL
* Thyroid stimulating hormone (TSH) within normal limits or thyroid disease under control
* Reconfirmation and documentation that sexually active female patients of childbearing potential are practicing adequate contraception (intrauterine device, oral contraceptives, progesterone implanted rods (Norplant), medroxyprogesterone acetate (Depo-Provera), surgical sterilization, barrier method (diaphragm + spermicide), or monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide) during the treatment period and for 6 months after discontinuation of therapy. A urine pregnancy test obtained at entry prior to the initiation of treatment must be negative. Female patients must not be breast-feeding. Documentation that sexually active male patients are practicing acceptable methods of contraception (vasectomy, use of a condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 6 months after discontinuation of therapy.
* Written informed consent specific for this protocol has been obtained prior to entry.

Exclusion Criteria:

* Hypersensitivity to interferon or ribavirin.
* Any cause for chronic liver disease other than chronic hepatitis C.
* Active hemolytic anemia.
* Evidence of advanced liver disease such as a history of or presence of ascites, bleeding varices, or spontaneous encephalopathy.
* Any known preexisting medical condition that could interfere with the patient's participation in the protocol including: (Central Nervous System) CNS trauma or uncontrolled seizure disorders; poorly controlled diabetes mellitus; serious pulmonary disease; immunologically-mediated diseases; gout' or any medical condition requiring, or likely to require during the course of the study, chronic administration of steroids.
* Patients with evidence of ischemia or stress testing, Electrocardiogram (ECG) evidence of ischemia, a significant arrhythmia, cardiac failure, recent coronary surgery, uncontrolled hypertension, angina or a myocardial infarction within 12 months. Pretreatment stress test will be required for all participants greater than 50 years of age or 45 years of age if diabetic.
* Patients with clinically significant retinal abnormalities.
* Substance abuse, such as alcohol (greater than 80 gm/day), intravenous (IV) drugs and inhaled drugs. If the patient has a history of substance abuse, to be considered for inclusion into the protocol, the patient must have abstained from using the abused substance for at least 3 months.
* Patients with a history of organ transplantation will be excluded.
* Patients infected with human immunodeficiency virus.
* Preexisting psychiatric conditions; especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, active suicidal ideation and/or suicidal attempt are excluded. Patients with a history of mild depression may enter the protocol if they meet the following eligibility criterion and are monitored more intensively. Mild depression includes either situational depression for a limited period or depressive symptoms, which do not significantly interfere with the patient's work or daily functions. All patients will complete the Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a 20-item self-report scale designed to measure depressive symptomatology experienced during the week prior to the interview. The items are scored on a four-point scale (0-3), with the total score ranging from zero to 60. CES-D scores of 16-20 suggest minor depression, and scores greater than 20 suggest major depression. The score can be determined in real time. A score of 16 or higher should prompt further questioning and consideration of treatment or referral to psychiatry. Detailed follow-up of each patient may be individualized according to his/her need; this would usually include predetermined visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, male or female, African-Americans or Caucasians, age 18 or older. Serum positive for hepatitis C.
Sampling Method: Non-Probability Sample
Enrollment: 260
Dates: Start 2001-03

PRIMARY OUTCOMES:
Determine if there is a difference in interferon-induced signaling between patients that respond to therapy and those that do not. | Analysis.
Measure and compare the sustained virologic response to standard treatment for hepatitis C between African American (AA) and non AA patients. | Analysis.
Determine how human leukocyte antigen (HLA) class II-dependent immune regulation and T cell specificities affect differences in immune responses to hepatitis C (HCV) and response to therapy in African American (AA) patients compared to non AA patients. | Analysis.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arkansas, Little Rock, Arkansas
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee